CLINICAL TRIAL: NCT06116227
Title: Efficacy of Whole-Body Vibration Training on Thermal Burn Injury in Paediatrics: A Prospective Randomized Controlled Trial
Brief Title: Whole-Body Vibration Training On Thermal Burn Injury In Pediatrics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadaya Mosaad, PHD (Principal Investigator), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24112004
Record Dates: First submitted 2023-10-21; First posted 2023-11-03 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Burns
Keywords: Whole-Body Vibration Training; Thermal burn; Pediatrics.
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Whole Body Vibration Training plus conventional physical therapy exercise program (Experimental): 30 patients received whole body vibration training on a vibration platform for 12-15 minutes, 3 times per week, plus a traditional physical therapy exercise program in the form of a 60-minute supervised exercise program for 8 weeks.
  Interventions: Device: Whole Body Vibration Training Plus Conventional Physical Therapy Exercise Program.; Other: Conventional Physical Therapy Exercise Program.
- Group B: Conventional Physical Therapy Exercise Program. (Experimental): 30 patients will receive a traditional physical therapy program. The program consists of 60 minutes of supervised exercise stretching exercise to all involved joints followed by strengthening for affected muscles for 8 weeks.
  Interventions: Other: Conventional Physical Therapy Exercise Program.

INTERVENTIONS:
Device: Whole Body Vibration Training Plus Conventional Physical Therapy Exercise Program. — Patients in the study group will receive the traditional physical therapy program first, followed immediately by whole-body vibration training on the vibration platform (Power Plate International, Irvine, California, USA) at the same visit. The vibration frequency will be 30 Hz and the amplitude will be from 4 to 7 mm, with an increase of 1mm every two weeks. The WBV program was three sessions a week for eight weeks. WBV duration starts with 10 min in the 1st week and up to 25 min in the 8th week, with a regular increase of five minutes after every two successive weeks.
  Arms: Group A: Whole Body Vibration Training plus conventional physical therapy exercise program
Other: Conventional Physical Therapy Exercise Program. — The program will include 60 minutes of a supervised and individualized exercise program, including stretching exercises for the Calf and hamstring muscles, followed by strengthening exercises for hip, knee, ankle, and foot muscles, and scar management techniques to avoid scar or contracture formation.

SUMMARY:
60 Patients with partial and full thickness thermal burns of the lower limb and trunk will be indiscriminately assigned to study group Group A(Study group): 30 patients received whole body vibration training on a vibration platform 12-15 minutes, 5 times per week, plus traditional physical therapy exercise program in the form of 60 minutes supervised exercise program for 8 weeks.

Group B (control group):30 patients will receive a traditional physical therapy program. The program consists of 60 minutes of supervised stretching exercise to all involved joints followed by strengthening for affected muscles for 8 weeks.

DETAILED DESCRIPTION:
The sample of participants will be chosen from the pediatric burn population by random generator and allocated randomly into two groups by permuted block randomization. Group (A): 30 patients received whole body vibration training on a vibration platform, the frequency, amplitude, and duration utilized in this investigation will be as follows: frequency: 30-40 Hz, 2-4 mm of peak-to-peak vertical plate displacement, and exercise durations ranging from 12-15 minutes. Participants will perform 2 vibration exercises 5 times per week for 8 weeks. The first vibration exercise, a warm-up and familiarization set, will consist of sitting in a chair with both legs on the platform and performing one repetition, which will last 3 minutes. At the completion of the 3-minute warm-up set, participants will perform 3 sets of 3-minute semi-squats on the vibration platform. Vibration exercise time will be increased by 30 seconds each week, with 3 minutes of rest being given between repetitions. The participants will be barefooted and wear similar cotton socks for each vibration session. Maintaining an upright body position, stand on their forefoot with their heels off the ground and the knee joints flexed at an angle of 10u. Their head and eyes were forward and distributed their weight equally on both feet with a foot-to-foot distance of 42 cm. Plus traditional physical therapy exercise programs in 60-minute supervised exercise programs.

Group (B): 30 patients will receive a traditional physical therapy program. The program consists of 60 minutes of supervised stretching exercise to all involved joints followed by strengthening for affected muscles for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age will range from 10 to 16 years
2. Patients of both sexes.
3. Participants have 25-40 % partial and full thickness burn of the lower limb and trunk.
4. Participants with complete wound healing or after 35-58 days from the start day of the injury.

Exclusion Criteria:

1. Patients with open burn wounds in any area of the body.
2. Patients diagnosed with acute rheumatoid arthritis
3. Diabetes, neuropathy, and neurological disorders.
4. Severe behavioral cognitive disorders.
5. Previous brain injury or any disease affecting balance, vestibular or visual disorders.
6. Patients with a history of traumatic spine within the past six months.
7. Patients with a prosthesis, Leg amputation, lower limb deformity, recent fracture or bone disease.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Balance Control: | 2 momths
  Biodex balance scale (Biodex medical systems Inc, Shirley, New York, USA), will be used for balance assessment that include overall stability index that is used to assess fluctuations around the zero point representing standard deviations rather than around a group mean. The overall stability index measures the fluctuations from the horizontal along axes of the Biodex stability system.

SECONDARY OUTCOMES:
Postural Stability | 2 months.
  The Berg balance scale includes 14 items with scores from 0 to 4. A score of 0 represents the inability to do the task, while a score of 4 represents the ability to do the task completely, according to the assigned criteria, with 56 indicates the total score. Items range from tasks of simple mobility(e.g. transfers, standing unsupported, sit-to-stand) to tasks with greater difficulty (e.g. tandem standing, turning 360°, single-leg stance).
Functional Mobility | 2 months.
  Timed-up and go test will be used. The test asks the participant to raise up from the sitting position followed by walking for 3 m, turning around, sitting again on the chair with his back supported, and resting his arms on the armrests.
Muscle Strength | 2 months.
  Muscle strength of the quadriceps and hamstring muscles will be assessed using a Biodex System-3 dynamometer (Biodex Medical System, Shirley, NY) prior to and following the 8-weeks intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadaya Mosaad Eladl, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
After 6 months of Publication, we can share the study protocol and Informed Consent form.
Supporting Information: Study Protocol, ICF
Time Frame: 6 months of Publication.